CLINICAL TRIAL: NCT04563533
Title: Phase I/IIa Clinical Trial to Evaluate the Safety, Tolerability and Immunogenicity of Longkoma Quadrivalent Recombinant Norovirus Vaccine (Pichia Pastoris) Implanted in Populations of 6 Weeks and Older
Brief Title: Clinical Trial of Quadrivalent Recombinant Norovirus Vaccine (Pichia Pastoris)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LKM-2020-NoV01
Record Dates: First submitted 2020-08-28; First posted 2020-09-24 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Acute Gastroenteritis
Keywords: prevention
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Intervention Model Description: A single-center, randomized, blinded, multi-cohort, placebo-controlled trial design was adopted.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subjects, investigators, monitors, and data analysts are not aware of treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- adults of phase I (Experimental): Healthy people aged 18-59
  Interventions: Biological: Low-dose vaccine; Biological: High-dose vaccine; Biological: Placebo (containing aluminum)
- teenagers of phase I (Experimental): Healthy people aged 6-17
  Interventions: Biological: Low-dose vaccine; Biological: High-dose vaccine; Biological: Placebo (containing aluminum)
- elderly of phase I (Placebo Comparator): Healthy people 60 years old and above
  Interventions: Biological: Low-dose vaccine; Biological: High-dose vaccine; Biological: Placebo (containing aluminum); Biological: Placebo (without aluminum)
- Toddler of phase I (Experimental): Healthy people aged 2-5
  Interventions: Biological: Low-dose vaccine; Biological: High-dose vaccine; Biological: Placebo (containing aluminum)
- Infants of phase I (Placebo Comparator): 6 weeks old-2 years old healthy person
  Interventions: Biological: Low-dose vaccine; Biological: High-dose vaccine; Biological: Placebo (containing aluminum); Biological: Placebo (without aluminum)
- elderly of phase II (Experimental): Healthy people 60 years old and above
  Interventions: Biological: Low-dose vaccine; Biological: High-dose vaccine
- Toddler of phase II (Placebo Comparator): Healthy people aged 2-5
  Interventions: Biological: Low-dose vaccine; Biological: High-dose vaccine
- Infants of phase II (Experimental): 6 weeks old-2 years old healthy person
  Interventions: Biological: Low-dose vaccine; Biological: High-dose vaccine

INTERVENTIONS:
Biological: Low-dose vaccine — Active ingredients: recombinant ReNoV GI.1-VP1 protein, recombinant ReNoV GII.3-VP1 protein, recombinant ReNoV GII.4-VP1 protein and recombinant ReNoV GII.17-VP1 protein each 12.5μg.
  Other ingredients: aluminum hydroxide adjuvant 0.25 mg, L-histidine: 1.55 mg, sodium chloride: 4 mg, Tween 80: 1 μg, sodium dihydrogen phosphate: 47 μg, disodium hydrogen phosphate: 87 μg.
Biological: High-dose vaccine — Active ingredients: recombinant ReNoV GI.1-VP1 protein, recombinant ReNoV GII.3-VP1 protein, recombinant ReNoV GII.4-VP1 protein and recombinant ReNoV GII.17-VP1 protein each 25μg.
  Other ingredients: aluminum hydroxide adjuvant 0.25 mg, L-histidine: 1.55 mg, sodium chloride: 4 mg, Tween 80: 2 μg, sodium dihydrogen phosphate: 94 μg, disodium hydrogen phosphate: 173 μg.
Biological: Placebo (containing aluminum) — Active ingredients: none Other ingredients: aluminum hydroxide adjuvant: 0.25 mg, L-histidine: 1.55 mg, sodium chloride: 4 mg, Tween 80: 2 μg, sodium dihydrogen phosphate: 94 μg, disodium hydrogen phosphate: 173 μg.
  Arms: Infants of phase I; Toddler of phase I; adults of phase I; elderly of phase I; teenagers of phase I
Biological: Placebo (without aluminum) — Active ingredients: none Other ingredients: L-histidine: 1.55 mg, sodium chloride: 4 mg, Tween 80: 2 μg, sodium dihydrogen phosphate: 94 μg, disodium hydrogen phosphate: 173 μg.
  Arms: Infants of phase I; elderly of phase I

SUMMARY:
The purpose of the research is to evaluate the safety and tolerability of the tetravalent recombinant Norovirus vaccine at different doses, to initially explore the immunogenicity of the vaccine, and to determine the appropriate dose of the product for later clinical trials.This trial adopts the seamless design of phase I/IIa, which is carried out in two phases, phase I and phase IIa, phase I is the age/dose climbing phase, and phase IIa is the dose expansion phase.It is planned to enroll 580 subjects, divided into 5 age groups, including: young adults (18-59 years old, 60 people), adolescents (6 -17 years old, 60 people), and elderly (≥60 years old, 160 people) , Toddlers (2-5 years old, 140), infants (6 weeks to 23 months old, 160).The test vaccine contains recombinant HuNoV GI.1-VP1 protein, HuNoV GII.3-VP1 protein, HuNoV GII.4-VP1 protein, HuNoV GII.17-VP1 protein, and each dose contains 12.5μg/type/0.5ml/bottle (Low dose), 25μg/type/0.5ml/piece (high dose).

DETAILED DESCRIPTION:
A single-center, randomized, blinded, multi-cohort, placebo-controlled trial design was adopted.This trial adopts the seamless design of phase I/IIa, which is carried out in two phases, phase I and phase IIa, phase I is the age/dose climbing phase, and phase IIa is the dose expansion phase.It is planned to enroll 580 subjects, divided into 5 age groups, including: young adults (18-59 years old, 60 people), adolescents (6 -17 years old, 60 people), and elderly (≥60 years old, 160 people) , Toddlers (2-5 years old, 140), infants (6 weeks to 23 months old, 160).Research phase and trial grouping: age/dose climbing phase: 340 subjects are planned to be enrolled in Liuzhou City, and they will be enrolled in the group according to the age order of young adults → adolescents and old people → toddlers → infants and young children. There are 10 cohorts, randomly divided into experimental group (low-dose or high-dose), placebo group (containing aluminum), and the random ratio of each entry stage is 2:1. Among them, infants and the elderly will be added a placebo group without aluminum adjuvant, test group (low dose or high dose), placebo group (aluminum), placebo (aluminum-free), the random ratio is 2:1:1; Dose expansion stage: It is planned to enroll 240 subjects in Rong'an County. The elderly, infants, and infants will be divided into 3 cohorts, and each age group will be randomly divided into low-dose or high-dose groups, with a random ratio of 1:1.According to the order of young adults → adolescents and elderly → toddlers → infants and young children, the dose is from low to high, and the investigator (including the main investigator and the field investigator) will review the safety of the low-dose/placebo group 7 days after the first dose. After the safety data is confirmed, you can enter the high-dose/placebo group for this age group to explore. After DSMB examines the safety data of the first dose of young and middle-aged people to 30 days after the full exemption and confirms safety, they can enter the adolescent and elderly age group; DSMB examines the safety and confirms the safety of the first dose of adolescents and the elderly to 30 days after the full exemption After that, you can enter the infant age group; the investigator (including the main investigator and the field investigator) will review the safety data 7 days after the first dose of the infant low-dose/placebo group and confirm the safety, then you can enter the infant age group explore. The three age groups (cohorts 4 and 6, 7 and 8, 9 and 10) of the elderly, toddlers, and infants can be entered into the corresponding age after the DSMB reviews the safety data of the first dose to 30 days after the full exemption and confirms the safety. In the dose expansion phase (cohorts 11, 12, 13), 80 subjects were enrolled in each cohort (of which, 40 were vaccinated with low-dose trial vaccine and 40 were vaccinated with high-dose trial vaccine).

ELIGIBILITY:
Inclusion Criteria:

1. Compliance with this clinical trial observation age is 6 weeks old and above, and can provide legal identification;
2. The suspected and/or violating legal guardian has the ability to understand the research procedures and sign an informed consent form;
3. Correct and/or prevent the legal guardian who has the ability to read, understand, fill in the diary card/contact card, and promise to participate regularly in accordance with the research requirements;
4. The armpit body temperature of all people on the day of entry was <37.3℃;
5. Standards for some groups of people:<12 months of age: singleton full-term pregnancy (37-42 weeks gestational week) and birth weight 2.5-4.0kg; women of childbearing age: agree to take effective contraceptive measures within 6 months after the first dose is implanted to the full exemption.

Exclusion Criteria:

1. The population laboratory test indicators specified in the plan are abnormal and have clinical significance;
2. A history of severe allergies to any component of the test vaccine, including L-histidine, sodium chloride, aluminum hydroxide, such as: anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergies Necrotic reaction (Arthus reaction); or any previous history of severe side effects of vaccines or drugs, such as: allergies, urticaria, skin eczema, dyspnea, angioedema, etc.;
3. 3 days before vaccination, suffering from acute disease or in the acute attack of chronic disease (such as asthma, diabetes, thyroid disease, etc.);
4. Have taken antipyretic or analgesics within 24 hours before the first dose of vaccination;
5. Inoculate the inactivated vaccine within 7 days before the first dose of vaccine, and the live attenuated vaccine within 14 days;
6. People suffering from the following diseases:①Suffered from digestive system diseases (such as diarrhea, abdominal pain, vomiting, etc.) in the past 7 days;② Suffer from severe congenital malformations, severe developmental disorders, severe genetic defects, severe malnutrition, etc.;③ Suffering from thrombocytopenia, any coagulation disorders or receiving anticoagulant treatment and other intramuscular injection contraindications;④ Congenital or acquired immunodeficiency, or receive immunosuppressive therapy within 6 months (for example, systemic glucocorticoid prednisone or similar drugs have been used for more than 2 consecutive weeks within 6 months). Local medications (such as ointments, eye drops, inhalants or nasal sprays) should not exceed the recommended dose in the instructions or show any signs of systemic exposure;⑤ Has been diagnosed with infectious diseases, such as tuberculosis, viral hepatitis and/or human immunodeficiency virus (HIV) infection;⑥ Having convulsions, epilepsy, encephalopathy (such as congenital brain hypoplasia, brain trauma, brain tumor, cerebral hemorrhage, cerebral obstruction, infection, chemical drug poisoning, etc. caused brain nerve tissue damage, etc.) and a history of mental illness or family history;⑦ No spleen, functional asthenia, as well as any cause of asthenia or splenectomy;⑧ Suffering from severe cardiovascular disease (pulmonary heart disease, pulmonary edema), severe liver and kidney disease, diabetes with complications;
7. Have received blood or blood-related products, including immunoglobulins, within 3 months, or plan to use them during the study period (within 1 month after enrollment and full exemption);
8. Any research or unregistered products (drugs, vaccines, biological products or devices) have been used within 3 months before enrollment, or planned to be used during the research period;
9. Plan to move or leave the local area for a long time during the research period;
10. Any situation that the researcher believes may interfere with the evaluation of the research purpose;
11. Standards for certain groups of people:①<12 months old: IVF, multiple fetuses, currently suffering from perianal abscess, severe eczema, pathological jaundice, parents with HIV infection;② Persons ≥18 years of age: Physical examination before enrollment is hypertension (systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg) or hypotension (systolic blood pressure <89mmHg) (regardless of medication);③Women of childbearing age: are breast-feeding or pregnant (including a positive urine pregnancy test) or have a pregnancy plan during the study period (in the group to within 6 months after the full exemption).

Min Age: 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
The number of adverse events after intramuscular injection | 6 months after full vaccination
  The main observation methods of adverse reactions mainly include laboratory examination, local reactions and systemic reactions at the administration site.
The positive conversion rate of norovirus antibody 30 days after the whole course of vaccination | 30 days after full immunization
  For young adults, the elderly, young children, infants and young children, the 4-fold growth rate of norovirus IgA, IgG, and HBGA blocking antibodies and the positive conversion rate after immunity were analyzed 30 days after the full immunization.

CONTACTS AND LOCATIONS:
Overall Officials: teng huang, master, Principal Investigator — Deputy Director of Vaccine Clinical Research Institute
Locations (1):
- Liuzhou Center for Disease Control and Prevention, Liuchow, Guangxi, China